CLINICAL TRIAL: NCT04173208
Title: Main Trial of the Cesarean Section and Intestinal Flora of the Newborn Study
Acronym: MT-SECFLOR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Helsinki (Other)
Responsible Party: Principal Investigator, Otto Helve, Adjunct professor, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT-SECFLOR
Record Dates: First submitted 2019-04-25; First posted 2019-11-21 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Fecal Microbiota Transplantation; Cesarean Section, Affecting Fetus or Newborn; Intestinal Microbiome
Keywords: Transplant; Cesarean section; inflammatory response; Infant

STUDY DESIGN:
Intervention Model Description: Number of enrolled mothers describes the number of mothers included for screening.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fecal microbial transplant (Experimental): The participants of the experimental arm will receive an oral fecal microbial transplant after delivery
  Interventions: Other: Fecal microbial transplant
- Placebo group (Placebo Comparator): The participants of the placebo arm will receive an oral placebo after delivery
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Fecal microbial transplant — Fecal microbial transplant
  Arms: Fecal microbial transplant
Other: Placebo — Placebo
  Arms: Placebo group

SUMMARY:
In this study the investigators assess whether, in CS-delivered infants, the intestinal microbiome could be successfully and safely normalised by postnatal oral transfer of maternal fecal microbiome.

DETAILED DESCRIPTION:
In this study the investigators assess whether, in CS-delivered infants, the intestinal microbiome could be successfully and safely normalised by postnatal oral transfer of maternal fecal microbiome. After faecal microbiota transfer, the children are followed for 24 months for the evaluation of markers of, for example, atopy-related diseases, and changes in immunomarkers associated with the transfer.

ELIGIBILITY:
Inclusion Criteria:

* non-eventful pregnancy
* planned elective CS
* Finnish language competency

Exclusion Criteria:

Mother:

* maternal refusal
* positive findings in screening samples
* maternal antibiotic treatment within 4 weeks of delivery (excluding the antibiotic given immediately prior to clamping of the umbilical cord)
* travel outside European Union during 3 months prior to delivery
* CS after the onset of labor (non-elective CS)

Newborn:

* birth below 37 weeks of gestation
* Apgar score of less than 8
* disturbances of neonatal adaptation (such as transient tachypnea of the newborn)
* antibiotic treatment of the newborn before discharge

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnancy
Enrollment: 90 (Actual)
Dates: Start 2019-11-10 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Longitudinal change of intestinal microbiota assessed with 16S rRNA and shotgun sequencing | At three months of age
  Developmental trajectory of the intestinal microbiota, assessed with 16s rRNA gene amplicon and shotgun sequencing of fecal DNA to determine the changes in the intestinal microbiota composition, diversity and functionality from birth to three months of age

SECONDARY OUTCOMES:
Difference in markers of cow milk immunoglobulin Es | At 12 months of age
  The difference in markers of allergen-specific immunoglobulin Es between the intervention group and the placebo group.
Difference in markers of aeroallergen immunoglobulin Es | At 24 months of age
  The difference in markers of allergen-specific immunoglobulin Es between the intervention group and the placebo group.
Difference in tetanus and measles, mumps and rubella vaccine responses | At 12 and 24 months of age
  The difference in vaccine responses between the intervention group and the placebo group (as Immunoglobulin G milli-International Units/milliliter).
Longitudinal change of intestinal microbiota assessed with 16S rRNA and shotgun sequencing | At 6, 12 and 24 months of age
  Developmental trajectory of the intestinal microbiota, assessed with 16s rRNA gene amplicon and shotgun sequencing of fecal DNA to determine the changes in the intestinal microbiota composition, diversity and functionality from birth to three months of age

OTHER OUTCOMES:
Differences in immunoresponse to the transplant | At 3 days and 3, 6, 12 and 24 months of age
  The differences in immunomarkers between the intervention group and the placebo group (measured by performing messenger ribonucleic acid sequencing of viable peripheral blood mononuclear cells).

CONTACTS AND LOCATIONS:
Overall Officials: Otto Helve, MD, PhD, Principal Investigator — Children's Hospital, Helsinki University Hospital and the University of Helsinki
Locations (1):
- Children's Hospital, Helsinki University Hospital, Pediatric Research Center, Helsinki, Uusimaa, Finland

REFERENCES:
- [Derived] Carpen N, Brodin P, de Vos WM, Salonen A, Kolho KL, Andersson S, Helve O. Transplantation of maternal intestinal flora to the newborn after elective cesarean section (SECFLOR): study protocol for a double blinded randomized controlled trial. BMC Pediatr. 2022 Sep 29;22(1):565. doi: 10.1186/s12887-022-03609-3. PMID 36175995